CLINICAL TRIAL: NCT05533996
Title: Body Fat Index as a Novel Sonographic Tool to Predict High Risk Pregnancy (BFiORS Trial)
Brief Title: Body Fat Index for Obstetric Risk Stratification
Acronym: BFIors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: Baylor College of Medicine (Other); Middle-Eastern College of Obstetricians and Gynecologists (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, Principal Investigator, The Leeds Teaching Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCOG-RCT02
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Gestational Diabetes; Pre-Eclampsia; Labour Dystocia
MeSH Terms: conditions — Diabetes, Gestational; Pre-Eclampsia | interventions — Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women prior to 14 weeks (Other): The sonographic examination will be conducted as an additional part after completing anatomical survey. . For the most accurate measurements, we will reduce the image depth to decrease the margin of error. We will conduct an initial abdominal sweep in all participants from the xiphoid to the umbilicus to detect the area of maximum pre-peritoneal fat thickness. Then, we will measure the maximum pre-peritoneal fat thickness and minimum subcutaneous fat thickness.
  Furthermore, all measurements will be conducted after inspiration to avoid its generated tension with the transducer just touching the skin avoiding compression of the subcutaneous fat. Two measurements will be taken to investigate the inter-observer effect. Then, BFI will be calculated using the following formula: BFI = pre-peritoneal fat (mm) x subcutaneous fat (mm) / Height (cm). Results will be communicated to the site primary investigator. The treating obstetrician will be blinded to these results.
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — Sonographic examination to measure the maternal pre-peritoneal fat thickness and subcutaneous fat thickness and calculate body fat index

SUMMARY:
Primary Outcome:- GDM Diagnosis Secondary Outcomes:- Pre-eclampsia diagnosis. Cesarean section delivery due to labor dystocia defined as protracted or arrested progress of labor using labor partogram.

DETAILED DESCRIPTION:
Obesity is one of the most common global risk factors for significant health issues, that has become increasingly prevalent among reproductive aged women. In the United States, obesity affects 21% in prepregnant females . Maternal obesity and excessive gestational weight gain have been linked to various adverse obstetric and neonatal outcomes, including spontaneous abortion, gestational diabetes mellitus (GDM), cesarean delivery, preeclampsia, neonatal macrosomia, and complications from surgery and anesthesia .

Consequently, contemporary guidelines recommend assessment of body mass index (BMI) at the first prenatal visit to guide diet and exercise directions and stratify obstetric risks . Nevertheless, BMI is associated with limitations to its clinical significance: first, it does not accurately correlate with the body fat distribution and does not differentiate between the increased mass of body muscle, bone, or fat being dependent on the patient's height and weight . Although all pregnant women with obesity is considered at risk of developing an adverse pregnancy outcome , women with BMI > 30 kg/m2 do not necessarily develop adverse outcomes, while women with BMI < 30 can still develop significant complications . Therefore, BMI does not present a clinically sensitive tool to screen and predict obesity-relevant adverse outcomes of pregnancy, including GDM, metabolic syndrome, and pre-eclampsia .

Anthropometric measurements such as waist circumference, hip circumference, waist/hip ratio, and others have been used to indicate that central fat is associated with the obesity-related adverse outcomes of pregnancy ; however, they are undermined by the subcutaneous fat amount . Computerized tomography (CT) and dual-energy X-ray absorptiometry have been implemented to measure visceral fat in the general population, which is deemed clinically related to health hazards. However, these approaches are associated with radiation exposure, associated with high costs, and are overall not appropriate for screening .

Ultrasound is safe during pregnancy and is routinely used as a part of antenatal care. Ultrasound can be used to measure visceral fat with similar sensitivity to CT in measuring fat thickness . Body fat index (BFI) is a novel tool that is calculated using the following formula (BFI = pre-peritoneal fat (mm) x subcutaneous fat (mm) / Height (cm)) . BFI was reported to be a safe, cost-effective, and easy screening method to identify the obesity-related adverse outcomes of pregnancy . Being dependent on pre-peritoneal fat which was reported to correlate with GDM with a predictive advantage over waist circumference and BMI , BFI constitutes a promising screening tool that can assess obesity-related adverse outcomes of pregnancy during first trimester scan without extra-costs and with high patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women prior to 14 weeks

Exclusion Criteria:

* Known pre-gestational diabetes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 206 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of gestational diabetes (GDM) | Between 24 and 28 weeks of pregnancy
  Diagnosis of GDM is made by abnormal glucose tolerance test during pregnancy

SECONDARY OUTCOMES:
Diagnosis of pre-eclampsia Incidence of Cesarean section | 24 weeks of pregnancy to 10 days postpartum
  The diagnosis is made by elevated blood pressure above 140 (systolic) and/or 90 (diastolic) in association with proteinuria
Labor dystocia | At time of labour (onset of labour pain to time of delivery)
  Failure to progress in labour resulting in Cesarean section delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Shazly, MSc, Principal Investigator — The Leeds Teaching Hospitals NHS Trust; Ahmed Nassr, MD, Principal Investigator — Baylor College of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaillard R, Durmus B, Hofman A, Mackenbach JP, Steegers EA, Jaddoe VW. Risk factors and outcomes of maternal obesity and excessive weight gain during pregnancy. Obesity (Silver Spring). 2013 May;21(5):1046-55. doi: 10.1002/oby.20088. PMID 23784909
- [Background] Haugen M, Brantsaeter AL, Winkvist A, Lissner L, Alexander J, Oftedal B, Magnus P, Meltzer HM. Associations of pre-pregnancy body mass index and gestational weight gain with pregnancy outcome and postpartum weight retention: a prospective observational cohort study. BMC Pregnancy Childbirth. 2014 Jun 11;14:201. doi: 10.1186/1471-2393-14-201. PMID 24917037
- [Background] Simon A, Pratt M, Hutton B, Skidmore B, Fakhraei R, Rybak N, Corsi DJ, Walker M, Velez MP, Smith GN, Gaudet LM. Guidelines for the management of pregnant women with obesity: A systematic review. Obes Rev. 2020 Mar;21(3):e12972. doi: 10.1111/obr.12972. Epub 2020 Jan 14. PMID 31943650
- [Background] Lee YS, Biddle S, Chan MF, Cheng A, Cheong M, Chong YS, Foo LL, Lee CH, Lim SC, Ong WS, Pang J, Pasupathy S, Sloan R, Seow M, Soon G, Tan B, Tan TC, Teo SL, Tham KW, van Dam RM, Wang J. Health Promotion Board-Ministry of Health Clinical Practice Guidelines: Obesity. Singapore Med J. 2016 Aug;57(8):472. doi: 10.11622/smedj.2016141. No abstract available. PMID 27550044
- [Background] ACOG Practice Bulletin No 156: Obesity in Pregnancy. Obstet Gynecol. 2015 Dec;126(6):e112-e126. doi: 10.1097/AOG.0000000000001211. No abstract available. PMID 26595582
- [Background] Fitzsimons KJ, Modder J; Centre for Maternal and Child Enquires. Setting maternity care standards for women with obesity in pregnancy. Semin Fetal Neonatal Med. 2010 Apr;15(2):100-7. doi: 10.1016/j.siny.2009.09.004. Epub 2009 Nov 25. PMID 19939755
- [Background] CDC. Body mass index: Considerations for practitioners. Cdc [Internet]. 2011;4.
- [Background] Heslehurst N, Ngongalah L, Bigirumurame T, Nguyen G, Odeniyi A, Flynn A, Smith V, Crowe L, Skidmore B, Gaudet L, Simon A, Hayes L. Association between maternal adiposity measures and adverse maternal outcomes of pregnancy: Systematic review and meta-analysis. Obes Rev. 2022 Jul;23(7):e13449. doi: 10.1111/obr.13449. Epub 2022 Apr 25. PMID 35467075
- [Background] Torloni MR, Betran AP, Horta BL, Nakamura MU, Atallah AN, Moron AF, Valente O. Prepregnancy BMI and the risk of gestational diabetes: a systematic review of the literature with meta-analysis. Obes Rev. 2009 Mar;10(2):194-203. doi: 10.1111/j.1467-789X.2008.00541.x. Epub 2008 Nov 24. PMID 19055539
- [Background] Roberts JM, Bodnar LM, Patrick TE, Powers RW. The Role of Obesity in Preeclampsia. Pregnancy Hypertens. 2011 Jan 1;1(1):6-16. doi: 10.1016/j.preghy.2010.10.013. PMID 21532964
- [Background] Chatzi L, Plana E, Daraki V, Karakosta P, Alegkakis D, Tsatsanis C, Kafatos A, Koutis A, Kogevinas M. Metabolic syndrome in early pregnancy and risk of preterm birth. Am J Epidemiol. 2009 Oct 1;170(7):829-36. doi: 10.1093/aje/kwp211. Epub 2009 Aug 27. PMID 19713286
- [Background] Gur EB, Ince O, Turan GA, Karadeniz M, Tatar S, Celik E, Yalcin M, Guclu S. Ultrasonographic visceral fat thickness in the first trimester can predict metabolic syndrome and gestational diabetes mellitus. Endocrine. 2014 Nov;47(2):478-84. doi: 10.1007/s12020-013-0154-1. Epub 2014 Jan 23. PMID 24452873
- [Background] Lukaski HC, Siders WA, Nielsen EJ, Hall CB. Total body water in pregnancy: assessment by using bioelectrical impedance. Am J Clin Nutr. 1994 Mar;59(3):578-85. doi: 10.1093/ajcn/59.3.578. PMID 8116533
- [Background] Bray GA, Jablonski KA, Fujimoto WY, Barrett-Connor E, Haffner S, Hanson RL, Hill JO, Hubbard V, Kriska A, Stamm E, Pi-Sunyer FX; Diabetes Prevention Program Research Group. Relation of central adiposity and body mass index to the development of diabetes in the Diabetes Prevention Program. Am J Clin Nutr. 2008 May;87(5):1212-8. doi: 10.1093/ajcn/87.5.1212. PMID 18469241
- [Background] Nassr AA, Shazly SA, Trinidad MC, El-Nashar SA, Marroquin AM, Brost BC. Body fat index: A novel alternative to body mass index for prediction of gestational diabetes and hypertensive disorders in pregnancy. Eur J Obstet Gynecol Reprod Biol. 2018 Sep;228:243-248. doi: 10.1016/j.ejogrb.2018.07.001. Epub 2018 Jul 6. PMID 30014931